CLINICAL TRIAL: NCT01618396
Title: Effects of Sedatives on Sublingual Microcirculation of Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa de Saúde São José (Other)
Responsible Party: Principal Investigator, Guilherme Loures Penna, Principal Investigator, Casa de Saúde São José
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CSSJ001
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Shock,; Sepsis
Keywords: Microcirculation; Hypnotics and Sedatives,; Propofol,; Midazolam
MeSH Terms: conditions — Shock; Sepsis | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sedation drug (Propofol and Midazolam) — Septic patients, after intubation, were initially sedated with propofol. During the second day of mechanical ventilation, propofol infusion was interrupted. When the patient awoke, the sedative drug was changed to midazolam. Sedation target was a Ramsay Scale score of 4 to 5.

SUMMARY:
Previous studies have demonstrated that altered microvascular blood flow is an important marker of severe sepsis. Usually, these patients need invasive ventilatory support, frequent use of sedatives and it is unknown if these agents interfere or not on microvascular blood flow. The goal of this study was to compare effects of propofol and midazolam infusions on sublingual microcirculation of septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients needing mechanical ventilation in pressure or volume-controlled mode.

Exclusion Criteria:

* age less than 18 years,
* pregnancy,
* non-sinus rhythm, and
* contraindication of daily interruption of sedative drug,
* mainly with the use of neuromuscular blocking drugs, or
* patients with intracranial hypertension or epileptical status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sublingual Microcirculatory Variables | Just before stopping propofol and thirty minutes after the start of midazolam infusion
  Patients were sedated with propofol during the first 24 hours after intubation and with midazolam afterwards.Systemic hemodynamics and perfusion parameters were assessed at two time points: just before stopping propofol and thirty minutes after the start of midazolam infusion. At both steps, four microcirculatory sequences were acquired using sidestream darkfield imaging to access sublingual microcirculation

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Penna, MD, MsC, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- Casa de Saude Sao Jose, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104. doi: 10.1164/rccm.200109-016oc. PMID 12091178
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Koch M, De Backer D, Vincent JL, Barvais L, Hennart D, Schmartz D. Effects of propofol on human microcirculation. Br J Anaesth. 2008 Oct;101(4):473-8. doi: 10.1093/bja/aen210. Epub 2008 Jul 23. PMID 18653494